CLINICAL TRIAL: NCT01390818
Title: An Open-Label, Phase Ib Dose Escalation Trial of Oral Combination Therapy With MSC1936369B and SAR245409 in Subjects With Locally Advanced or Metastatic Solid Tumors
Brief Title: Trial of MEK Inhibitor and PI3K/mTOR Inhibitor in Subjects With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR 200066-006
Record Dates: First submitted 2011-04-18; First posted 2011-07-11 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2017-03-07 (Actual); Status verified 2017-01

CONDITIONS: Locally Advanced Solid Tumor; Metastatic Solid Tumor; Breast Cancer; Non Small Cell Lung Cancer; Melanoma; Colorectal Cancer
Keywords: MEK inhibitor (Pimasertib); PI3K/mTOR Inhibitor; Solid Tumor; Phase I
MeSH Terms: conditions — Neoplasm Metastasis; Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Melanoma; Colorectal Neoplasms | interventions — N-(2,3-dihydroxypropyl)-1-((2-fluoro-4-iodophenyl)amino)isonicotinamide; XL765; Phosphatidylinositol 3-Kinases; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MSC1936369B and SAR245409 once daily (Experimental)
  Interventions: Drug: MSC1936369B (pimasertib); Drug: SAR245409 (PI3K and mTOR inhibitor)
- MSC1936369B and SAR245409 twice daily (Experimental)
  Interventions: Drug: MSC1936369B (pimasertib); Drug: SAR245409 (PI3K and mTOR inhibitor)

INTERVENTIONS:
Drug: MSC1936369B (pimasertib) — MSC1936369B (pimasertib) single dose capsule was administered at dose of 15 milligram (mg), 30 mg, 60 mg, 90 mg orally in successive 21-day cycles.Dose escalation was proceeded until Maximum Tolerated Dose (MTD) was reached. Once the MTD was reached, enrollment began in four disease-specific expansion cohorts at either the MTD or a lower dose recommended by the Safety Monitoring Committee. The four expansion cohorts enrolled subjects with Breast Cancer, Non-Small Cell Lung Cancer (NSCLC), Melanoma, and Colorectal Cancer.
  Other Names: Pimasertib
  Arms: MSC1936369B and SAR245409 once daily
Drug: SAR245409 (PI3K and mTOR inhibitor) — SAR245409 (PI3K and mTOR inhibitor) capsule was administered orally at a dose of 30 mg, 50 mg, 70 mg and 90 mg in successive 21-day cycles. Dose escalation was proceeded until MTD was reached. Once the MTD was reached, enrollment began in four disease-specific expansion cohorts at either the MTD or a lower dose recommended by the Safety Monitoring Committee. The four expansion cohort enrolled subjects with Breast Cancer, NSCLC, Melanoma, and Colorectal Cancer.
  Other Names: PI3K and mTOR inhibitor
  Arms: MSC1936369B and SAR245409 once daily
Drug: MSC1936369B (pimasertib) — MSC1936369B (pimasertib) capsule was administered twice daily orally at a dose of 60 mg and 45 mg in successive 21-day cycles. Dose escalation proceeded until MTD was reached. The maximum tolerated dose of MSC1936369B (pimasertib) was combined with a lower dose of SAR245409 (PI3K and mTOR inhibitor).
  Other Names: pimasertib
  Arms: MSC1936369B and SAR245409 twice daily
Drug: SAR245409 (PI3K and mTOR inhibitor) — SAR245409 (PI3K and mTOR inhibitor) was administered twice daily orally at a dose of 30 mg and 50 mg in successive 21-day cycles. Dose escalation proceeded until MTD was reached. The maximum tolerated dose of SAR245409 (PI3K and mTOR inhibitor) was combined with a lower dose of MSC1936369B (pimasertib).
  Other Names: PI3K and mTOR inhibitor
  Arms: MSC1936369B and SAR245409 twice daily

SUMMARY:
This research trial is testing a combination of two experimental drugs, MSC1936369B (Mitogen-activated protein extracellular signal-regulated kinase (MEK) Inhibitor) and SAR245409 (Phosphatidylinositol 3-kinase (Pi3K)/Mammalian Target of Rapamycin (mTOR) inhibitor), in the treatment of locally advanced or metastatic solid tumors. The primary purpose of the study is to determine the maximum tolerated dose of the drug combination.

ELIGIBILITY:
Inclusion Criteria:

* Subject with advanced solid tumors for which there is no approved therapy:

  * Advanced solid tumor with diagnosed alteration in one or more of the following genes (PTEN, BRAF, KRAS, NRAS, PI3KCA, ErbB1, ErbB2, MET, RET, c-KIT, GNAQ, GNA11 and/or
  * A histologically or cytologically confirmed diagnosis of one of the following solid tumors: pancreatic, thyroid, colorectal, non-small cell lung, endometrial, renal, breast, ovarian carcinoma and melanoma
* Subject with archived tumor tissue available for transfer to the Sponsor
* Subject enrolled at lower dose level cohorts and MTD expansion cohorts must have tumor available for biopsy and agree to pre-treatment and on-treatment tumor biopsies
* Subject has measurable or evaluable disease by response evaluation criteria in solid tumors (RECIST) v1.1
* Subject is aged greater than or equal to (>=) 18 years
* Subjects enrolled in disease specific expansion cohorts must fulfill all the inclusion/exclusion criteria listed above with the following restriction to the Inclusion Criterion number 1:

  * Relapsed or refractory Kirsten rat sarcoma viral oncogene homolog (KRAS) or neuroblastoma RAS viral oncogene homolog (NRAS) mutated metastatic non-small cell lung cancer (NSCLC) with no approved therapies, or
  * Relapsed or refractory metastatic triple negative breast cancer defined as estrogen, progesterone and HER2 negative carcinoma of the breast with no approved therapies, or
  * Relapsed or refractory metastatic colorectal cancer (CRC) with dual KRAS and PIK3CA mutation with no approved therapies, or
  * BRAF V600E/K mutated unresectable or metastatic melanoma after progression on B-Raf proto-oncogene, serine/threonine kinase (BRAF) inhibitors
* Other protocol-defined inclusion criteria could apply

Exclusion Criteria:

* Subject has been previously treated with a PI3K inhibitor or a MEK inhibitor and taken off treatment due to treatment related adverse events
* Subject has received:
* Chemotherapy, immunotherapy, hormonal therapy, biologic therapy, or any other anti-cancer therapy within 28 days of trial drug treatment
* Any investigational agent within 28 days of trial drug treatment
* Extensive prior radiotherapy on more than 30% bone marrow reserves, or prior bone marrow/stem cell transplantation
* Subject has not recovered from toxicity due to prior therapy
* Subject has poor organ and marrow function as defined in the protocol
* Subject has a history of central nervous system metastases, unless subject has been previously treated for CNS metastases
* Subject has a history of difficulty swallowing, malabsorption or other chronic gastrointestinal disease
* Subject has a history of recent major surgery or trauma within the last 28 days.
* Subject has participated in another clinical trial within the past 30 days
* Other protocol-defined exclusion criteria could apply

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2011-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono, a business of Merck KGaA, Darmstadt, Germany
Locations (8):
- United States (6):
  - Pinnacle Oncology Hematology, Scottsdale, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Cancer Therapy and Research Center, San Antonio, Texas
- Merck Serono Research Site, Milan, Italy
- Merck Serono Research Site, Madrid, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject (informed consent): May 2011. Study completion date: Apr 2015. A total of 192 subjects were screened and 146 subjects entered the trial and received the investigational medicinal product (IMP).
Pre-assignment Details: Study had a 4-day Drug-Drug Interaction (DDI) period, within 1 week prior to Day 1 Cycle 1, to assess possible interaction only in selected subjects where in SAR245409 and Pimasertib were administered alone on Day 1 and Day 3, respectively.
Groups:
- Pimasertib (MSC1936369B) 15mg and SAR245409 30mg Once Daily: Pimasertib (MSC1936369B) capsule was administered at a single oral dose of 15 milligram (mg) along with single oral dose of 30 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (Dose Escalation [DE] cohort).
- Pimasertib (MSC1936369B) 30mg and SAR245409 30mg Once Daily: Pimasertib (MSC1936369B) capsule was administered at a single oral dose of 30 mg along with single oral dose of 30 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- Pimasertib (MSC1936369B) 15mg and SAR245409 50mg Once Daily: Pimasertib (MSC1936369B) capsule was administered at a single oral dose of 15 mg along with single oral dose of 50 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- Pimasertib (MSC1936369B) 30mg and SAR245409 50mg Once Daily: Pimasertib (MSC1936369B) capsule was administered at a single oral dose of 30 mg along with single oral dose of 50 mg SAR245409 capsule on Day 1 of each 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- Pimasertib (MSC1936369B) 60mg and SAR245409 50mg Once Daily: Pimasertib (MSC1936369B) capsule was administered at a single oral dose of 60 mg along with single oral dose of 50 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- Pimasertib (MSC1936369B) 30mg and SAR245409 70mg Once Daily: Pimasertib (MSC1936369B) capsule was administered at a single oral dose of 30 mg along with single oral dose of 70 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- Pimasertib (MSC1936369B) 60mg and SAR245409 70mg Once Daily: Pimasertib (MSC1936369B) capsule was administered at a single oral dose of 60 mg along with single oral dose of 70 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- Pimasertib (MSC1936369B) 90mg and SAR245409 70mg Once Daily: Pimasertib (MSC1936369B) capsule was administered at a single oral dose of 90 mg along with single oral dose of 70 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- Pimasertib (MSC1936369B) 60mg and SAR245409 90mg Once Daily: Pimasertib (MSC1936369B) capsule was administered at a single oral dose of 60 mg along with single oral dose of 90 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- Pimasertib (MSC1936369B) 60mg and SAR245409 30mg Twice Daily: Pimasertib (MSC1936369B) capsule was administered twice orally at a dose of 60 mg along with twice oral dose of 30 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- Pimasertib (MSC1936369B) 45mg and SAR245409 50mg Twice Daily: Pimasertib (MSC1936369B) capsule was administered twice orally at a dose of 45 mg along with twice oral dose of 50 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- TNBC: Pimasertib 60mg and SAR245409 70mg Once Daily: Subjects with relapsed or refractory metastatic triple negative breast cancer (TNBC) defined as estrogen, progesterone, and human epidermal growth factor receptor 2 (HER2) negative carcinoma of the breast with no approved therapies in disease specific expansion (DSE) cohort received Pimasertib (MSC1936369B) capsule at a single oral dose of 60 mg along with single oral dose of 70 mg SAR245409 capsule on Day 1 of each 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject.
- NSCLC: Pimasertib 60mg and SAR245409 70mg Once Daily: Subjects with a histologically confirmed diagnosis of relapsed or refractory metastatic non-small cell lung cancer (NSCLC) in disease specific expansion (DSE) cohort received Pimasertib (MSC1936369B) capsule at a single oral dose of 60 mg along with single oral dose of 70 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject.
- CRC: Pimasertib 60mg and SAR245409 70mg Once Daily: Subjects with relapsed or refractory metastatic colorectal carcinoma/cancer (CRC) in DSE cohort received Pimasertib (MSC1936369B) capsule at a single oral dose of 60 mg along with single oral dose of 70 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject.
- MEL: Pimasertib 60mg and SAR245409 70mg Once Daily: Subjects with relapsed or refractory metastatic melanoma (MEL) in DSE cohort received Pimasertib (MSC1936369B) capsule at a single oral dose of 60 mg along with single oral dose of 70 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject.
Period: Overall Study
Arm/Group | Pimasertib (MSC1936369B) 15mg and SAR245409 30mg Once Daily | Pimasertib (MSC1936369B) 30mg and SAR245409 30mg Once Daily | Pimasertib (MSC1936369B) 15mg and SAR245409 50mg Once Daily | Pimasertib (MSC1936369B) 30mg and SAR245409 50mg Once Daily | Pimasertib (MSC1936369B) 60mg and SAR245409 50mg Once Daily | Pimasertib (MSC1936369B) 30mg and SAR245409 70mg Once Daily | Pimasertib (MSC1936369B) 60mg and SAR245409 70mg Once Daily | Pimasertib (MSC1936369B) 90mg and SAR245409 70mg Once Daily | Pimasertib (MSC1936369B) 60mg and SAR245409 90mg Once Daily | Pimasertib (MSC1936369B) 60mg and SAR245409 30mg Twice Daily | Pimasertib (MSC1936369B) 45mg and SAR245409 50mg Twice Daily | TNBC: Pimasertib 60mg and SAR245409 70mg Once Daily | NSCLC: Pimasertib 60mg and SAR245409 70mg Once Daily | CRC: Pimasertib 60mg and SAR245409 70mg Once Daily | MEL: Pimasertib 60mg and SAR245409 70mg Once Daily
Started | 3 | 3 | 3 | 4 | 4 | 3 | 19 | 14 | 3 | 3 | 4 | 26 | 24 | 18 | 15
Completed | 3 | 3 | 3 | 4 | 4 | 3 | 19 | 14 | 3 | 3 | 4 | 26 | 24 | 18 | 15
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety analysis set (SAF) included subjects who received at least one (non-zero) administration of the trial IMPs (pimasertib and/or SAR245409).
Groups:
- Pimasertib (MSC1936369B) 15mg and SAR245409 30mg Once Daily: Pimasertib (MSC1936369B) capsule was administered at a single oral dose of 15 milligram (mg) along with single oral dose of 30 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- Pimasertib (MSC1936369B) 30mg and SAR245409 50mg Once Daily: Pimasertib (MSC1936369B) capsule was administered at a single oral dose of 30 mg along with single oral dose of 50 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- Total: Total of all reporting groups
Arm/Group | Pimasertib (MSC1936369B) 15mg and SAR245409 30mg Once Daily | Pimasertib (MSC1936369B) 30mg and SAR245409 30mg Once Daily | Pimasertib (MSC1936369B) 15mg and SAR245409 50mg Once Daily | Pimasertib (MSC1936369B) 30mg and SAR245409 50mg Once Daily | Pimasertib (MSC1936369B) 60mg and SAR245409 50mg Once Daily | Pimasertib (MSC1936369B) 30mg and SAR245409 70mg Once Daily | Pimasertib (MSC1936369B) 60mg and SAR245409 70mg Once Daily | Pimasertib (MSC1936369B) 90mg and SAR245409 70mg Once Daily | Pimasertib (MSC1936369B) 60mg and SAR245409 90mg Once Daily | Pimasertib (MSC1936369B) 60mg and SAR245409 30mg Twice Daily | Pimasertib (MSC1936369B) 45mg and SAR245409 50mg Twice Daily | TNBC: Pimasertib 60mg and SAR245409 70mg Once Daily | NSCLC: Pimasertib 60mg and SAR245409 70mg Once Daily | CRC: Pimasertib 60mg and SAR245409 70mg Once Daily | MEL: Pimasertib 60mg and SAR245409 70mg Once Daily | Total
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 4 | 3 | 19 | 14 | 3 | 3 | 4 | 26 | 24 | 18 | 15 | 146
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 1 | 2 | 1 | 2 | 16 | 12 | 3 | 2 | 2 | 22 | 16 | 12 | 13 | 107
  >=65 years | 1 | 2 | 2 | 2 | 3 | 1 | 3 | 2 | 0 | 1 | 2 | 4 | 8 | 6 | 2 | 39
Gender [Count of Participants; unit: Participants]
  Female | 3 | 1 | 2 | 1 | 1 | 1 | 6 | 13 | 1 | 2 | 0 | 26 | 15 | 11 | 4 | 87
  Male | 0 | 2 | 1 | 3 | 3 | 2 | 13 | 1 | 2 | 1 | 4 | 0 | 9 | 7 | 11 | 59

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Dose Limiting Toxicities (DLT)
Description: DLT was defined as any of the following toxicities experienced during the first cycle of treatment at any dose level (DL) and judged not to be related to the underlying disease or any concomitant medication by the Investigator and/or the Sponsor: A treatment emergent adverse event (TEAE) of potential clinical significance such that further dose escalation (DE) would have exposed subjects to unacceptable risk. Any Grade greater than or equal to (>=) 3 non-hematological toxicity, except for: Grade 3 diarrhea, nausea and vomiting with a duration less than or equal to (<=) 48 hours despite adequate supportive care and Alopecia. Grade 4 neutropenia of > 5 days duration or febrile neutropenia. Grade 3 thrombocytopenia with bleeding or Grade 4 thrombocytopenia. Any treatment interruption > 2 weeks due to AEs not related to the underlying disease or concomitant medication at any dose level and any severe, life-threatening impairing daily functions complication or abnormality.
Time Frame: Day 1 up to Day 16 in cycle 1
Population: The dose escalation (DE) analysis set included all subjects treated in DE cohorts who received at least 80 percent (%) of pimasertib and 80% of SAR245409 full planned doses in the first cycle (ie, 21-day period from Day 1) of treatment or who experienced a DLT during the first cycle of treatment regardless of the received amount of each drug.
Measure: Number; unit: subjects
Arm/Group | Pimasertib (MSC1936369B) 15mg and SAR245409 30mg Once Daily | Pimasertib (MSC1936369B) 30mg and SAR245409 30mg Once Daily | Pimasertib (MSC1936369B) 15mg and SAR245409 50mg Once Daily | Pimasertib (MSC1936369B) 30mg and SAR245409 50mg Once Daily | Pimasertib (MSC1936369B) 60mg and SAR245409 50mg Once Daily | Pimasertib (MSC1936369B) 30mg and SAR245409 70mg Once Daily | Pimasertib (MSC1936369B) 60mg and SAR245409 70mg Once Daily | Pimasertib (MSC1936369B) 90mg and SAR245409 70mg Once Daily | Pimasertib (MSC1936369B) 60mg and SAR245409 90mg Once Daily | Pimasertib (MSC1936369B) 60mg and SAR245409 30mg Twice Daily | Pimasertib (MSC1936369B) 45mg and SAR245409 50mg Twice Daily
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 2 | 3 | 11 | 11 | 2 | 3 | 4
subjects | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 1

2. Secondary Outcome: Number of Subjects Experiencing Any Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a subject administered a pharmaceutical product, which did not necessarily have a causal relationship with this treatment. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAEs were defined as those AEs that started between first dose of study drug and up to 30 days after last dose.
Time Frame: Baseline up to 30 Days after last dose; assessed up to 4 years
Population: The safety analysis set (SAF) analysis set was to include all subjects who had received at least 1 (non-zero) administration of the trial investigational medicinal products (IMPs) MSC1936369B (pimasertib) and/or SAR245409.
Measure: Number; unit: subjects
Groups:
- Pimasertib (MSC1936369B) 15mg and SAR245409 30mg Once Daily: Pimasertib (MSC1936369B) capsule was administered at a single oral dose of 15 mg along with single oral dose of 30 mg SAR245409 capsule on Day 1 of each 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- Pimasertib (MSC1936369B) 30mg and SAR245409 30mg Once Daily: Pimasertib (MSC1936369B) capsule was administered at a single oral dose of 30 mg along with single oral dose of 30 mg SAR245409 capsule on Day 1 of each 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- Pimasertib (MSC1936369B) 15mg and SAR245409 50mg Once Daily: Pimasertib (MSC1936369B) capsule was administered at a single oral dose of 15 mg along with single oral dose of 50 mg SAR245409 capsule on Day 1 of each 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- Pimasertib (MSC1936369B) 60mg and SAR245409 50mg Once Daily: Pimasertib (MSC1936369B) capsule was administered at a single oral dose of 60 mg along with single oral dose of 50 mg SAR245409 capsule on Day 1 of each 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- Pimasertib (MSC1936369B) 30mg and SAR245409 70mg Once Daily: Pimasertib (MSC1936369B) capsule was administered at a single oral dose of 30 mg along with single oral dose of 70 mg SAR245409 capsule on Day 1 of each 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- Pimasertib (MSC1936369B) 60mg and SAR245409 70mg Once Daily: Pimasertib (MSC1936369B) capsule was administered at a single oral dose of 60 mg along with single oral dose of 70 mg SAR245409 capsule on Day 1 of each 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- Pimasertib (MSC1936369B) 90mg and SAR245409 70mg Once Daily: Pimasertib (MSC1936369B) capsule was administered at a single oral dose of 90 mg along with single oral dose of 70 mg SAR245409 capsule on Day 1 of each 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- Pimasertib (MSC1936369B) 60mg and SAR245409 90mg Once Daily: Pimasertib (MSC1936369B) capsule was administered at a single oral dose of 60 mg along with single oral dose of 90 mg SAR245409 capsule on Day 1 of each 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- MSC1936369B (Pimasertib) 45mg and SAR245409 50mg Twice Daily: Pimasertib (MSC1936369B) capsule was administered twice orally at a dose of 45 mg along with twice oral dose of 50 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- NSCLC: Pimasertib 60mg and SAR245409 70mg Once Daily: Subjects with a histologically confirmed diagnosis of relapsed or refractory metastatic non-small cell lung cancer (NSCLC) in disease specific expansion (DSE) cohort received Pimasertib (MSC1936369B) capsule at a single oral dose of 60 mg along with single oral dose of 70 mg SAR245409 capsule on Day 1 of each 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject.
- CRC: Pimasertib 60mg and SAR245409 70mg Once Daily: Subjects with relapsed or refractory metastatic colorectal carcinoma/cancer (CRC) in DSE cohort received Pimasertib (MSC1936369B) capsule at a single oral dose of 60 mg along with single oral dose of 70 mg SAR245409 capsule on Day 1 of each 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject.
- MEL: Pimasertib 60mg and SAR245409 70mg Once Daily: Subjects with relapsed or refractory metastatic melanoma (MEL) in DSE cohort received Pimasertib (MSC1936369B) capsule at a single oral dose of 60 mg along with single oral dose of 70 mg SAR245409 capsule on Day 1 of each 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject.
Arm/Group | Pimasertib (MSC1936369B) 15mg and SAR245409 30mg Once Daily | Pimasertib (MSC1936369B) 30mg and SAR245409 30mg Once Daily | Pimasertib (MSC1936369B) 15mg and SAR245409 50mg Once Daily | Pimasertib (MSC1936369B) 30mg and SAR245409 50mg Once Daily | Pimasertib (MSC1936369B) 60mg and SAR245409 50mg Once Daily | Pimasertib (MSC1936369B) 30mg and SAR245409 70mg Once Daily | Pimasertib (MSC1936369B) 60mg and SAR245409 70mg Once Daily | Pimasertib (MSC1936369B) 90mg and SAR245409 70mg Once Daily | Pimasertib (MSC1936369B) 60mg and SAR245409 90mg Once Daily | Pimasertib (MSC1936369B) 60mg and SAR245409 30mg Twice Daily | MSC1936369B (Pimasertib) 45mg and SAR245409 50mg Twice Daily | TNBC: Pimasertib 60mg and SAR245409 70mg Once Daily | NSCLC: Pimasertib 60mg and SAR245409 70mg Once Daily | CRC: Pimasertib 60mg and SAR245409 70mg Once Daily | MEL: Pimasertib 60mg and SAR245409 70mg Once Daily
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 4 | 3 | 19 | 14 | 3 | 3 | 4 | 26 | 24 | 18 | 15
subjects | 3 | 3 | 3 | 4 | 4 | 3 | 19 | 14 | 3 | 3 | 4 | 26 | 24 | 18 | 15

3. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Pimasertib (MSC1936369B)
Time Frame: Predose 0.5, 1, 1.5, 2, 3, 4, 8 and 24 hour post dose on Day 1, 15 for DSE Cohorts; Predose 0.5, 1, 1.5, 2, 3, 4, 8, 10 and 24 hour post dose on Day 1, 15 for DE cohorts
Population: The pharmacokinetic (PK) analysis set. Here "n" signifies the number of subjects evaluable at the specific time points.
Measure: Geometric Mean (95% Confidence Interval); unit: nanogram/millilitre (ng/mL)
Groups:
- Pimasertib (MSC1936369B) 15mg: Pimasertib (MSC1936369B) capsule administered at a single oral dose of 15 milligram (mg) on Day 1 of 21 day cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- Pimasertib (MSC1936369B) 30mg: Pimasertib (MSC1936369B) capsule administered at a single oral dose of 30 mg on Day 1 of 21 day cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- Pimasertib (MSC1936369B) 60mg: Pimasertib (MSC1936369B) capsule administered at a single oral dose of 60 mg on Day 1 of 21 day cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- Pimasertib (MSC1936369B) 90mg: Pimasertib (MSC1936369B) capsule administered at a single oral dose of 90 mg on Day 1 and 15 of cycle 1 until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- Pimasertib (MSC1936369B) 45mg Twice Daily: Pimasertib (MSC1936369B) capsule administered twice, orally, at a dose of 45 mg on Day 1 and 15 of cycle 1 until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- Pimasertib (MSC1936369B) 60mg Twice Daily: Pimasertib (MSC1936369B) capsule administered twice, orally, at a dose of 60 mg on Day 1 and 15 of cycle 1 until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- TNBC: Pimasertib 60mg Once Daily; NSCLC: Pimasertib 60mg Once Daily; CRC: Pimasertib 60mg Once Daily; MEL: Pimasertib 60mg Once Daily: Pimasertib (MSC1936369B) capsule administered at a single oral dose of 60 mg on Day 1 and 15 of cycle 1 until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DSE Cohort).
Arm/Group | Pimasertib (MSC1936369B) 15mg | Pimasertib (MSC1936369B) 30mg | Pimasertib (MSC1936369B) 60mg | Pimasertib (MSC1936369B) 90mg | Pimasertib (MSC1936369B) 45mg Twice Daily | Pimasertib (MSC1936369B) 60mg Twice Daily | TNBC: Pimasertib 60mg Once Daily | NSCLC: Pimasertib 60mg Once Daily | CRC: Pimasertib 60mg Once Daily | MEL: Pimasertib 60mg Once Daily
Number analyzed (Participants) | 6 | 10 | 26 | 14 | 4 | 3 | 26 | 24 | 18 | 15
nanogram/millilitre (ng/mL)
  Day 1 (n=6, 10, 26, 13, 4, 3, 25, 23, 18, 15) | 86.06 [51.31 to 144.3] | 188.2 [138.5 to 255.9] | 246.1 [191.8 to 315.6] | 406.9 [284.6 to 581.7] | 83.72 [18.05 to 388.3] | 232.5 [190.9 to 283.2] | 323.1 [253.9 to 411.1] | 295.4 [240.9 to 362.2] | 245.6 [198.5 to 304.0] | 234.0 [182.6 to 299.8]
  Day 15 (n=6, 9,15,9, 3, 1, 16, 17, 13, 10) | 131.3 [85.13 to 202.6] | 212.8 [178.9 to 253.1] | 234.2 [166.2 to 330.1] | 516.4 [375.0 to 711.0] | 143.1 [22.82 to 897.8] | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 320.5 [286.2 to 358.9] | 327.6 [248.5 to 431.9] | 307.7 [205.0 to 461.8] | 338.9 [281.0 to 408.8]

4. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Pimasertib (MSC1936369B)
Time Frame: as for outcome 3
Population: The PK analysis set. Here "n" signifies the number of subjects evaluable at the specific time points.
Measure: Median (Full Range); unit: hour
Groups:
- Pimasertib (MSC1936369B) 90mg: Pimasertib (MSC1936369B) capsule administered at a single oral dose of 90 mg on Day 1 of 21 day cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- Pimasertib (MSC1936369B) 45mg Twice Daily: Pimasertib (MSC1936369B) capsule administered twice, orally, at a dose of 45 mg on Day 1 of 21 day cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- Pimasertib (MSC1936369B) 60mg Twice Daily: Pimasertib (MSC1936369B) capsule administered twice, orally, at a dose of 60 mg on Day 1 of 21 day cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE cohort).
- TNBC: Pimasertib 60mg Once Daily; NSCLC: Pimasertib 60mg Once Daily; CRC: Pimasertib 60mg Once Daily; MEL: Pimasertib 60mg Once Daily: Pimasertib (MSC1936369B) capsule administered at a single oral dose of 60 mg on Day 1 of 21 day cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DSE Cohort).
Arm/Group | Pimasertib (MSC1936369B) 15mg | Pimasertib (MSC1936369B) 30mg | Pimasertib (MSC1936369B) 60mg | Pimasertib (MSC1936369B) 90mg | Pimasertib (MSC1936369B) 45mg Twice Daily | Pimasertib (MSC1936369B) 60mg Twice Daily | TNBC: Pimasertib 60mg Once Daily | NSCLC: Pimasertib 60mg Once Daily | CRC: Pimasertib 60mg Once Daily | MEL: Pimasertib 60mg Once Daily
Number analyzed (Participants) | 6 | 10 | 26 | 14 | 4 | 3 | 26 | 24 | 18 | 15
hour
  Day 1 (n= 6, 10, 25, 13, 4, 3, 25, 23, 18, 15 ) | 1.750 [0.50 to 2.08] | 0.765 [0.50 to 2.15] | 2.020 [0.50 to 8.05] | 1.500 [0.50 to 3.00] | 1.485 [0.50 to 2.08] | 1.550 [0.50 to 2.07] | 1.500 [0.50 to 7.90] | 1.520 [0.50 to 7.85] | 1.490 [0.50 to 4.20] | 1.050 [0.45 to 4.00]
  Day 15 (n= 6, 9, 15, 9, 3, 1, 16, 17, 13, 10) | 1.275 [0.50 to 3.07] | 1.000 [1.00 to 1.63] | 2.000 [1.00 to 7.95] | 1.550 [1.00 to 2.00] | 2.000 [1.50 to 4.17] | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 1.505 [0.53 to 3.00] | 1.530 [1.00 to 4.00] | 1.500 [0.50 to 8.00] | 1.030 [0.48 to 3.83]

5. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) From Time Zero to the Last Sampling Time (0-24 Hours) of Pimasertib (MSC1936369B)
Description: Area under the concentration-time curve from time 0 to the last quantifiable concentration.
Time Frame: as for outcome 3
Population: The PK analysis set . Here "n" signifies the number of subjects evaluable at the specific time points.
Measure: Geometric Mean (95% Confidence Interval); unit: hour*nanogram per millilitre (hr*ng/mL)
Arm/Group | Pimasertib (MSC1936369B) 15mg | Pimasertib (MSC1936369B) 30mg | Pimasertib (MSC1936369B) 60mg | Pimasertib (MSC1936369B) 90mg | Pimasertib (MSC1936369B) 45mg Twice Daily | Pimasertib (MSC1936369B) 60mg Twice Daily | TNBC: Pimasertib 60mg Once Daily | NSCLC: Pimasertib 60mg Once Daily | CRC: Pimasertib 60mg Once Daily | MEL: Pimasertib 60mg Once Daily
Number analyzed (Participants) | 6 | 10 | 26 | 14 | 4 | 3 | 26 | 24 | 18 | 15
hour*nanogram per millilitre (hr*ng/mL)
  Day 1 (n=6, 10, 25, 13, 4, 3, 25, 23, 18, 15) | 426.8 [306.2 to 594.9] | 734.4 [586.1 to 920.3] | 1547 [1238 to 1934] | 2116 [1664 to 2692] | 326.1 [110.9 to 958.7] | 1252 [1100 to 1425] | 1781 [1404 to 2260] | 1754 [1480 to 2078] | 1709 [1361 to 2146] | 1093 [871.5 to 1371]
  Day 15 (n=6, 9,15,9, 3, 1, 16, 17, 10, 13) | 625.3 [405.7 to 963.9] | 902.0 [747.6 to 1088] | 1617 [1170 to 2236] | 2552 [2185 to 2980] | 773.1 [201.0 to 2974] | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 2136 [1713 to 2663] | 1889 [1540 to 2318] | 1988 [1487 to 2658] | 1506 [1141 to 1988]

6. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC 0-inf) of Pimasertib (MSC1936369B) at Day 1
Description: Area under the concentration-time curve from time 0 extrapolated to infinity, calculated as AUC0-t + last observed concentration (Clast)/terminal rate constant (λz), using the Linear up/Log down method.
  Terminal rate constant (λz).
Time Frame: Predose 0.5, 1, 1.5, 2, 3, 4, 8 and 24 hour post dose on Day 1 for DSE Cohorts; Predose 0.5, 1, 1.5, 2, 3, 4, 8, 10 and 24 hour post dose on Day 1 for DE cohorts
Population: The PK analysis set. Here "N" signifies the number of subjects evaluable for this outcome measure. Data was not available for 'Pimasertib (MSC1936369B) 60mg Twice Daily' arm as no subjects were considered evaluable because of limited number of samples collected to characterize the terminal phase rate constant needed for the calculation of AUCinf.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ng/mL
Arm/Group | Pimasertib (MSC1936369B) 15mg | Pimasertib (MSC1936369B) 30mg | Pimasertib (MSC1936369B) 60mg | Pimasertib (MSC1936369B) 90mg | Pimasertib (MSC1936369B) 45mg Twice Daily | Pimasertib (MSC1936369B) 60mg Twice Daily | TNBC: Pimasertib 60mg Once Daily | NSCLC: Pimasertib 60mg Once Daily | CRC: Pimasertib 60mg Once Daily | MEL: Pimasertib 60mg Once Daily
Number analyzed (Participants) | 6 | 9 | 23 | 13 | 3 | 0 | 22 | 22 | 14 | 13
hr*ng/mL | 451.6 [319.8 to 637.8] | 770.9 [599.9 to 990.6] | 1607 [1237 to 2087] | 2202 [1716 to 2826] | 503.1 [153.1 to 1654] |  | 1869 [1451 to 2407] | 1830 [1518 to 2207] | 1857 [1414 to 2437] | 1113 [858.9 to 1442]

7. Secondary Outcome: Area Under the Concentration-Time Curve (AUC) During a Dosing Interval (Tau) of Pimasertib (MSC1936369B)
Time Frame: as for outcome 3
Population: The PK analysis set. Here "n" signifies the number of subjects evaluable at the specific time points.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ng/mL
Arm/Group | Pimasertib (MSC1936369B) 15mg | Pimasertib (MSC1936369B) 30mg | Pimasertib (MSC1936369B) 60mg | Pimasertib (MSC1936369B) 90mg | Pimasertib (MSC1936369B) 45mg Twice Daily | Pimasertib (MSC1936369B) 60mg Twice Daily | TNBC: Pimasertib 60mg Once Daily | NSCLC: Pimasertib 60mg Once Daily | CRC: Pimasertib 60mg Once Daily | MEL: Pimasertib 60mg Once Daily
Number analyzed (Participants) | 6 | 10 | 26 | 14 | 4 | 3 | 26 | 24 | 18 | 15
hr*ng/mL
  Day 1 (n= 6, 10, 26, 13, 3, 3, 24, 23, 17,13) | 426.8 [306.2 to 594.9] | 742.1 [602.0 to 914.7] | 1547 [1238 to 1934] | 2116 [1664 to 2692] | 354.9 [48.21 to 2613] | 1252 [1100 to 1425] | 1882 [1513 to 2341] | 1754 [1480 to 2078] | 1772 [1409 to 2227] | 1093 [871.5 to 1371]
  Day 15 (n=6, 9, 15, 9, 3, 0, 16, 17, 10, 13) | 650.4 [440.1 to 961.2] | 902.0 [747.6 to 1088] | 1617 [1170 to 2236] | 2552 [2185 to 2980] | 773.1 [201.0 to 2974] | NA [NA to NA] — Data could not be calculated because there were no subjects evaluated for this arm at the specified time point. | 2136 [1713 to 2663] | 1889 [1540 to 2318] | 1988 [1487 to 2658] | 1506 [1141 to 1988]

8. Secondary Outcome: Half-Life (t1/2) of MSC1936369B (Pimasertib)
Time Frame: as for outcome 3
Population: The PK analysis set. Here "n" signifies the number of subjects evaluable at the specific time points.
Measure: Median (Full Range); unit: hour
Arm/Group | Pimasertib (MSC1936369B) 15mg | Pimasertib (MSC1936369B) 30mg | Pimasertib (MSC1936369B) 60mg | Pimasertib (MSC1936369B) 90mg | Pimasertib (MSC1936369B) 45mg Twice Daily | Pimasertib (MSC1936369B) 60mg Twice Daily | TNBC: Pimasertib 60mg Once Daily | NSCLC: Pimasertib 60mg Once Daily | CRC: Pimasertib 60mg Once Daily | MEL: Pimasertib 60mg Once Daily
Number analyzed (Participants) | 6 | 10 | 26 | 14 | 4 | 3 | 26 | 24 | 18 | 15
hour
  Day 1 (n=6, 9, 23, 13, 4, 3, 22, 22, 15, 13) | 6.250 [5.03 to 7.16] | 4.670 [1.85 to 5.79] | 4.840 [3.23 to 9.99] | 4.800 [3.49 to 7.62] | 3.320 [2.60 to 4.72] | 4.640 [4.25 to 4.74] | 4.840 [2.46 to 8.41] | 4.370 [3.71 to 8.26] | 4.770 [3.51 to 12.8] | 4.240 [3.32 to 4.84]
  Day 15 (n=6, 9, 14, 9, 2, 1, 16, 16, 9, 12) | 5.855 [2.93 to 7.88] | 5.410 [3.90 to 10.8] | 6.755 [4.61 to 14.3] | 5.590 [3.97 to 14.1] | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 5.210 [3.25 to 12.8] | 5.250 [4.33 to 8.65] | 5.210 [4.80 to 6.94] | 4.325 [3.40 to 5.96]

9. Secondary Outcome: Total Body Clearance (CL/f) of Pimasertib (MSC1936369B)
Description: The total body clearance of drug from plasma following oral administration (Cl/f) and the total body clearance of drug from plasma following intravenous administration was calculated by dividing the Dose with area under the plasma concentration time curve from time zero to infinity (AUC0 inf)=Dose/AUC0- inf.
Time Frame: as for outcome 3
Population: The PK analysis set. Here "N" signifies number of subjects evaluable for this outcome measure and "n" signifies the number of subjects evaluable at the specific time points.
Measure: Geometric Mean (95% Confidence Interval); unit: litre per hour (L/hr)
Arm/Group | Pimasertib (MSC1936369B) 15mg | Pimasertib (MSC1936369B) 30mg | Pimasertib (MSC1936369B) 60mg | Pimasertib (MSC1936369B) 90mg | Pimasertib (MSC1936369B) 45mg Twice Daily | Pimasertib (MSC1936369B) 60mg Twice Daily | TNBC: Pimasertib 60mg Once Daily | NSCLC: Pimasertib 60mg Once Daily | CRC: Pimasertib 60mg Once Daily | MEL: Pimasertib 60mg Once Daily
Number analyzed (Participants) | 6 | 10 | 26 | 14 | 4 | 1 | 26 | 24 | 18 | 15
litre per hour (L/hr)
  Day 1 (n=6, 10, 26, 13, 3, 0, 22, 22, 14, 13) | 33.22 [23.52 to 46.92] | 38.90 [30.26 to 50.00] | 37.99 [29.33 to 49.22] | 40.88 [31.85 to 52.47] | 89.49 [27.14 to 295.1] | NA [NA to NA] — Data could not be calculated because there were no subjects evaluated for this arm at the specified time point. | 32.12 [24.95 to 41.36] | 32.75 [27.16 to 39.50] | 30.75 [23.41 to 40.41] | 53.94 [41.61 to 69.62]
  Day 15 (n=6, 9, 15, 9, 3, 1, 16, 17, 10, 13) | 23.06 [15.59 to 34.10] | 33.30 [27.63 to 40.13] | 37.11 [26.82 to 51.33] | 35.28 [30.19 to 41.23] | 58.22 [15.03 to 225.6] | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 28.11 [22.54 to 35.07] | 31.73 [25.85 to 38.94] | 30.20 [22.59 to 40.38] | 39.81 [30.17 to 52.52]

10. Secondary Outcome: Apparent Volume of Distribution of Total Pimasertib During the Terminal Phase Following Oral Administration (Vz/f) of Pimasertib
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/f) was influenced by the fraction absorbed. Apparent volume of distribution during the terminal phase, calculated by CL/f/λz. Terminal rate constant (λz). The regression analysis (determination of λz) was to contain as many data points as possible (but excluding Cmax) and had to include concentration data from at least 3 different time points, consistent with the assessment of a straight line (the terminal elimination phase) on the log-transformed scale.Data was not available for 'Pimasertib (MSC1936369B) 60mg Twice Daily' arm as no subjects were considered evaluable because of limited number of samples collected to characterize the terminal phase rate constant needed for the calculation of Vz/f.
Time Frame: as for outcome 3
Population: The PK analysis set. Here "N" signifies number of subjects evaluable for this outcome measure and "n" signifies the number of subjects evaluable at specific time points.
Measure: Geometric Mean (95% Confidence Interval); unit: liter
Arm/Group | Pimasertib (MSC1936369B) 15mg | Pimasertib (MSC1936369B) 30mg | Pimasertib (MSC1936369B) 60mg | Pimasertib (MSC1936369B) 90mg | Pimasertib (MSC1936369B) 45mg Twice Daily | Pimasertib (MSC1936369B) 60mg Twice Daily | TNBC: Pimasertib 60mg Once Daily | NSCLC: Pimasertib 60mg Once Daily | CRC: Pimasertib 60mg Once Daily | MEL: Pimasertib 60mg Once Daily
Number analyzed (Participants) | 6 | 10 | 26 | 14 | 3 | 0 | 26 | 24 | 18 | 15
liter
  Day 1 (n=6, 9, 23, 13, 3, 0, 22, 22, 14, 13) | 294.3 [218.5 to 396.4] | 240.2 [202.5 to 284.9] | 282.8 [227.7 to 351.4] | 283.0 [224.0 to 357.6] | 394.1 [146.9 to 1058] |  | 223.8 [182.7 to 274.3] | 226.9 [193.9 to 265.4] | 216.2 [174.6 to 267.8] | 322.0 [251.5 to 412.3]
  Day 15 (n=6, 9, 13, 9, 0, 0, 16, 16, 9, 12) | 188.7 [133.4 to 266.9] | 261.8 [187.9 to 364.8] | 396.4 [276.9 to 567.3] | 302.4 [223.1 to 409.7] | NA [NA to NA] — Data could not be calculated because there were no subjects evaluated for this arm at the specified time point because of limited number of samples collected to characterize the terminal phase rate constant needed for the calculation of Vz/f. |  | 226.3 [189.7 to 270.1] | 250.9 [214.2 to 293.9] | 230.6 [169.0 to 314.6] | 273.8 [213.8 to 350.7]

11. Secondary Outcome: Accumulation Ratio (Racc) for AUCtau of Pimasertib (MSC1936369B): Day 15
Description: Accumulation ratio (Racc) for AUCtau, calculated as Day 15 dosing interval AUCtau per Day 1 dosing interval AUCtau.
Time Frame: as for outcome 3
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Groups:
- Pimasertib (MSC1936369B) 15mg: Pimasertib (MSC1936369B) capsule administered at a single oral dose of 15 mg on Day 1 of 21 day cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE Cohort).
Arm/Group | Pimasertib (MSC1936369B) 15mg | Pimasertib (MSC1936369B) 30mg | Pimasertib (MSC1936369B) 60mg | Pimasertib (MSC1936369B) 90mg | Pimasertib (MSC1936369B) 45mg Twice Daily | Pimasertib (MSC1936369B) 60mg Twice Daily | TNBC: Pimasertib 60mg Once Daily | NSCLC: Pimasertib 60mg Once Daily | CRC: Pimasertib 60mg Once Daily | MEL: Pimasertib 60mg Once Daily
Number analyzed (Participants) | 6 | 9 | 15 | 9 | 3 | 1 | 15 | 17 | 10 | 13
ratio | 1.523 [1.295 to 1.792] | 1.269 [1.107 to 1.455] | 1.174 [0.9326 to 1.479] | 1.364 [1.133 to 1.642] | 2.176 [0.1184 to 39.99] | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 1.368 [1.044 to 1.792] | 1.155 [1.004 to 1.330] | 1.245 [0.9538 to 1.625] | 1.283 [1.104 to 1.490]

12. Secondary Outcome: Accumulation Ratio (Racc) for Cmax of Pimasertib (MSC1936369B): Day 15
Description: Accumulation ratio (Racc) for Cmax, calculated as Day 15 Cmax/Day 1 Cmax.
Time Frame: as for outcome 3
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Pimasertib (MSC1936369B) 15mg | Pimasertib (MSC1936369B) 30mg | Pimasertib (MSC1936369B) 60mg | Pimasertib (MSC1936369B) 90mg | Pimasertib (MSC1936369B) 45mg Twice Daily | Pimasertib (MSC1936369B) 60mg Twice Daily | TNBC: Pimasertib 60mg Once Daily | NSCLC: Pimasertib 60mg Once Daily | CRC: Pimasertib 60mg Once Daily | MEL: Pimasertib 60mg Once Daily
Number analyzed (Participants) | 6 | 9 | 15 | 9 | 3 | 1 | 16 | 17 | 10 | 13
ratio | 1.525 [1.002 to 2.322] | 1.066 [0.7442 to 1.527] | 1.106 [0.7904 to 1.546] | 1.308 [0.7537 to 2.268] | 1.467 [0.02541 to 84.67] | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 1.203 [0.9074 to 1.595] | 1.059 [0.8875 to 1.263] | 1.247 [0.8719 to 1.784] | 1.393 [1.091 to 1.780]

13. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for SAR245409
Time Frame: as for outcome 3
Population: The PK analysis set. Here "n" signifies the number of subjects evaluable at the specific time points.
Measure: Geometric Mean (95% Confidence Interval); unit: nanogram per millilitre (ng/mL)
Groups:
- SAR245409 30mg: SAR245409 capsule administered at a single oral dose of 30 milligram (mg) on Day 1 of 21 day cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE Cohort).
- SAR245409 50mg: SAR245409 capsule administered at a single oral dose of 50 mg on Day 1 of 21 day cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE Cohort).
- SAR245409 70mg: SAR245409 capsule administered at a single oral dose of 70 mg on Day 1 of 21 day cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE Cohort).
- SAR245409 90mg: SAR245409 capsule administered at a single oral dose of 90 mg on Day 1 of 21 day cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE Cohort).
- SAR245409 30mg Twice Daily: SAR245409 capsule administered twice, orally, at a dose of 30 mg on Day 1 of 21 day cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE Cohort).
- SAR245409 50mg Twice Daily: SAR245409 capsule administered twice, orally, at a dose of 50 mg on Day 1 of 21 day cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DE Cohort).
- TNBC: SAR245409 70mg Once Daily; NSCLC: SAR245409 70mg Once; CRC: SAR245409 70mg Once Daily; MEL: SAR245409 70mg Once Daily: SAR245409 capsule administered at a single oral dose of 70 mg on Day 1 of 21 day cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DSE Cohort).
Arm/Group | SAR245409 30mg | SAR245409 50mg | SAR245409 70mg | SAR245409 90mg | SAR245409 30mg Twice Daily | SAR245409 50mg Twice Daily | TNBC: SAR245409 70mg Once Daily | NSCLC: SAR245409 70mg Once | CRC: SAR245409 70mg Once Daily | MEL: SAR245409 70mg Once Daily
Number analyzed (Participants) | 6 | 11 | 36 | 3 | 3 | 4 | 26 | 24 | 18 | 15
nanogram per millilitre (ng/mL)
  Day 1 (n=6, 11, 36, 3, 3, 4, 26, 23, 18, 15) | 192.0 [115.6 to 316.3] | 295.7 [189.0 to 462.6] | 256.9 [203.5 to 324.3] | 224.5 [99.72 to 505.2] | 130.2 [20.76 to 816.5] | 64.22 [19.25 to 214.2] | 323.6 [258.4 to 405.2] | 240.6 [164.6 to 351.6] | 239.6 [158.8 to 361.4] | 212.5 [129.3 to 349.4]
  Day 15 (n=6, 6, 25, 1, 1, 3, 17, 17, 10, 13) | 199.8 [114.4 to 349.1] | 224.1 [132.7 to 378.4] | 222.9 [143.7 to 345.7] | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 117.2 [7.210 to 1907] | 326.0 [256.4 to 414.6] | 235.5 [144.6 to 383.3] | 178.9 [82.31 to 389.0] | 226.6 [143.9 to 356.7]

14. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of SAR245409
Description: The time to reach maximum plasma concentration (Tmax) of SAR245409 was calculated.
Time Frame: as for outcome 3
Population: The PK analysis set. Here "n" signifies the number of subjects evaluable at the specific time points.
Measure: Median (Full Range); unit: hours
Groups:
- NSCLC: SAR245409 70mg Once Daily; CRC: SAR245409 70mg Once Daily; MEL: SAR245409 70mg Once Daily: SAR245409 capsule administered at a single oral dose of 70 mg on Day 1 of 21 day cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DSE Cohort).
Arm/Group | SAR245409 30mg | SAR245409 50mg | SAR245409 70mg | SAR245409 90mg | SAR245409 30mg Twice Daily | SAR245409 50mg Twice Daily | TNBC: SAR245409 70mg Once Daily | NSCLC: SAR245409 70mg Once Daily | CRC: SAR245409 70mg Once Daily | MEL: SAR245409 70mg Once Daily
Number analyzed (Participants) | 6 | 11 | 36 | 3 | 3 | 4 | 26 | 24 | 18 | 15
hours
  Day 1 (n=6, 11, 36, 3, 3, 4, 26, 23, 18, 15) | 1.510 [0.53 to 2.08] | 1.150 [0.50 to 4.10] | 1.500 [0.50 to 23.80] | 1.500 [1.00 to 8.00] | 2.050 [1.50 to 2.07] | 1.540 [0.50 to 4.00] | 1.500 [0.52 to 8.03] | 2.000 [0.50 to 4.17] | 2.000 [0.43 to 8.05] | 1.500 [0.95 to 4.00]
  Day 15 (n=6, 8, 25, 1, 1, 3, 17, 17, 10, 13) | 1.265 [1.00 to 2.00] | 1.750 [0.53 to 3.00] | 1.970 [1.00 to 8.13] | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 1.550 [1.50 to 8.00] | 2.030 [0.52 to 7.98] | 1.530 [0.92 to 8.00] | 1.750 [0.50 to 8.00] | 1.050 [0.50 to 3.97]

15. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) From Time Zero to the Last Sampling Time (0-24 Hours) of SAR245409
Description: Area under the plasma concentration-time curve (AUC) from time zero to the last sampling time (0-24 hours) at which the concentration is at or above the lower limit of quantification. Unit of assessment was hour*nanogram per milliliter (hr*ng/mL).
Time Frame: as for outcome 3
Population: The PK analysis set. Here "n" signifies the number of subjects evaluable at the specific time points.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ng/mL
Arm/Group | SAR245409 30mg | SAR245409 50mg | SAR245409 70mg | SAR245409 90mg | SAR245409 30mg Twice Daily | SAR245409 50mg Twice Daily | TNBC: SAR245409 70mg Once Daily | NSCLC: SAR245409 70mg Once Daily | CRC: SAR245409 70mg Once Daily | MEL: SAR245409 70mg Once Daily
Number analyzed (Participants) | 6 | 11 | 36 | 3 | 3 | 4 | 26 | 24 | 18 | 15
hr*ng/mL
  Day 1 (n=6, 11, 36, 3, 3, 4, 26, 23, 18, 15) | 683.6 [248.9 to 1878] | 1248 [760.1 to 2050] | 1566 [1162 to 2111] | 3032 [1425 to 6454] | 634.0 [111.8 to 3595] | 226.2 [82.99 to 616.7] | 1976 [1449 to 2693] | 1408 [962.5 to 2059] | 1479 [824.6 to 2653] | 854.9 [505.0 to 1447]
  Day 15 (n=6, 8, 25, 1, 1, 3, 17, 17, 10, 13) | 861.0 [371.5 to 1995] | 1125 [558.3 to 2266] | 1334 [895.8 to 1986] | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 537.5 [56.10 to 5150] | 2232 [1512 to 3297] | 1437 [922.1 to 2239] | 1365 [543.4 to 3431] | 968.8 [554.8 to 1692]

16. Secondary Outcome: Area Under the Concentration-Time Curve (AUC) During a Dosing Interval (Tau) of SAR245409
Time Frame: as for outcome 3
Population: The PK analysis set. Here "n" signifies the number of subjects evaluable at the specific time points.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ng/mL
Arm/Group | SAR245409 30mg | SAR245409 50mg | SAR245409 70mg | SAR245409 90mg | SAR245409 30mg Twice Daily | SAR245409 50mg Twice Daily | TNBC: SAR245409 70mg Once Daily | NSCLC: SAR245409 70mg Once Daily | CRC: SAR245409 70mg Once Daily | MEL: SAR245409 70mg Once Daily
Number analyzed (Participants) | 6 | 11 | 36 | 3 | 3 | 4 | 26 | 24 | 18 | 15
hr*ng/mL
  Day 1 (n=6, 11, 36, 3, 3, 3, 24, 23, 17, 15) | 746.9 [275.5 to 2024] | 1265 [784.5 to 2041] | 1601 [1195 to 2145] | 3032 [1425 to 6454] | 634.0 [111.8 to 3595] | 298.6 [120.4 to 740.6] | 2115 [1535 to 2915] | 1480 [1026 to 2137] | 1542 [851.5 to 2792] | 948.4 [601.8 to 1495]
  Day 15 (n=6, 8, 25, 1, 1, 3, 17, 17, 10, 13) | 887.9 [397.9 to 1981] | 1168 [611.5 to 2232] | 1362 [918.9 to 2018] | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 537.5 [56.10 to 5150] | 2390 [1696 to 3368] | 1437 [922.1 to 2239] | 1365 [543.4 to 3431] | 1074 [636.9 to 1811]

17. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) From Time Zero to Infinity (0-inf) of SAR245409: Day 1
Description: Area under the concentration-time curve from time 0 extrapolated to infinity, calculated as AUC0-t + last observed concentration (Clast)/terminal rate constant (λz), using the Linear up/Log down method.
  Terminal rate constant (λz). The regression analysis (determination of λz) was to contain as many data points as possible (but excluding Cmax) and had to include concentration data from at least 3 different time points, consistent with the assessment of a straight line (the terminal elimination phase) on the log-transformed scale.
Time Frame: as for outcome 6
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ng/mL
Arm/Group | SAR245409 30mg | SAR245409 50mg | SAR245409 70mg | SAR245409 90mg | SAR245409 30mg Twice Daily | SAR245409 50mg Twice Daily | TNBC: SAR245409 70mg Once Daily | NSCLC: SAR245409 70mg Once Daily | CRC: SAR245409 70mg Once Daily | MEL: SAR245409 70mg Once Daily
Number analyzed (Participants) | 5 | 9 | 31 | 2 | 1 | 3 | 20 | 17 | 12 | 12
hr*ng/mL | 716.5 [181.8 to 2823] | 1165 [648.3 to 2093] | 1504 [1113 to 2034] | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 331.2 [151.5 to 724.1] | 1974 [1408 to 2768] | 1445 [1019 to 2049] | 1261 [579.4 to 2743] | 1142 [750.4 to 1739]

18. Secondary Outcome: Apparent Terminal Half-Life (t1/2) of SAR245409
Time Frame: as for outcome 3
Population: The PK analysis set. Here "n" signifies the number of subjects evaluable at the specific time points.
Measure: Median (Full Range); unit: hour
Arm/Group | SAR245409 30mg | SAR245409 50mg | SAR245409 70mg | SAR245409 90mg | SAR245409 30mg Twice Daily | SAR245409 50mg Twice Daily | TNBC: SAR245409 70mg Once Daily | NSCLC: SAR245409 70mg Once Daily | CRC: SAR245409 70mg Once Daily | MEL: SAR245409 70mg Once Daily
Number analyzed (Participants) | 6 | 11 | 36 | 3 | 3 | 4 | 26 | 24 | 18 | 15
hour
  Day 1 (n=6, 9, 31, 2, 2, 3, 20, 19, 13, 14) | 3.055 [1.78 to 7.57] | 3.300 [1.45 to 8.94] | 3.390 [0.964 to 9.28] | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 3.310 [2.47 to 3.37] | 3.755 [1.32 to 7.59] | 3.300 [2.54 to 27.9] | 4.070 [2.14 to 9.02] | 3.120 [1.32 to 6.03]
  Day 15 (n=6, 8, 22, 1, 1, 2, 10, 15, 8, 10) | 3.700 [2.07 to 5.60] | 4.570 [1.81 to 6.49] | 4.560 [2.37 to 35.2] | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 2.840 [1.48 to 5.63] | 4.050 [2.74 to 7.87] | 6.170 [3.43 to 11.8] | 3.065 [1.79 to 5.37]

19. Secondary Outcome: Total Body Clearance (CL/f) of SAR245409
Description: The total body clearance of drug from plasma following oral administration (Cl/f) and the total body clearance of drug from plasma following intravenous administration was calculated by dividing the dose with area under the plasma concentration time curve from time zero to infinity (AUC 0-inf)=Dose/AUC 0-inf.
Time Frame: as for outcome 3
Population: The PK analysis set. Here "n" signifies the number of subjects evaluable at the specific time points.
Measure: Geometric Mean (95% Confidence Interval); unit: litre per hour
Arm/Group | SAR245409 30mg | SAR245409 50mg | SAR245409 70mg | SAR245409 90mg | SAR245409 30mg Twice Daily | SAR245409 50mg Twice Daily | TNBC: SAR245409 70mg Once Daily | NSCLC: SAR245409 70mg Once Daily | CRC: SAR245409 70mg Once Daily | MEL: SAR245409 70mg Once Daily
Number analyzed (Participants) | 6 | 11 | 36 | 2 | 1 | 4 | 26 | 24 | 18 | 15
litre per hour
  Day 1 (n=5, 9, 31, 2, 1, 3, 20, 17, 12, 12) | 41.80 [10.62 to 164.5] | 42.93 [23.89 to 77.16] | 46.54 [34.42 to 62.94] | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 151.4 [69.37 to 330.4] | 35.43 [25.26 to 49.69] | 48.40 [34.12 to 68.64] | 55.51 [25.52 to 120.7] | 61.29 [40.26 to 93.30]
  Day 15 (n=6, 8, 25, 1, 1, 3, 17, 17, 10, 13) | 33.78 [15.16 to 75.26] | 42.81 [22.39 to 81.85] | 51.38 [34.68 to 76.13] | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 92.90 [9.667 to 892.8] | 29.28 [20.78 to 41.26] | 48.69 [31.25 to 75.88] | 51.24 [20.38 to 128.8] | 65.16 [38.64 to 109.9]

20. Secondary Outcome: Apparent Volume of Distribution of Total SAR245409 During the Terminal Phase Following Oral Administration (Vz/f)
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/f) was influenced by the fraction absorbed. Apparent volume of distribution during the terminal phase, calculated by CL/f/λz. Terminal rate constant (λz). The regression analysis (determination of λz) was to contain as many data points as possible (but excluding Cmax) and had to include concentration data from at least 3 different time points, consistent with the assessment of a straight line (the terminal elimination phase) on the log-transformed scale.
Time Frame: as for outcome 3
Population: The PK analysis set. Here "n" signifies the number of subjects evaluable at the specific time points.
Measure: Geometric Mean (95% Confidence Interval); unit: litre
Arm/Group | SAR245409 30mg | SAR245409 50mg | SAR245409 70mg | SAR245409 90mg | SAR245409 30mg Twice Daily | SAR245409 50mg Twice Daily | TNBC: SAR245409 70mg Once Daily | NSCLC: SAR245409 70mg Once Daily | CRC: SAR245409 70mg Once Daily | MEL: SAR245409 70mg Once Daily
Number analyzed (Participants) | 6 | 11 | 36 | 2 | 1 | 4 | 26 | 24 | 18 | 15
litre
  Day 1 (n=5, 9, 31, 2, 1, 3, 20, 17, 12, 12) | 174.8 [71.24 to 429.0] | 223.4 [116.2 to 429.6] | 238.5 [179.0 to 317.8] | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 658.0 [211.9 to 2044] | 175.2 [123.9 to 247.9] | 251.4 [158.4 to 398.9] | 353.6 [177.1 to 705.8] | 270.3 [175.6 to 416.0]
  Day 15 (n=6, 8, 25, 1, 1, 2, 17, 17, 10, 13 ) | 165.7 [99.48 to 276.1] | 257.2 [156.7 to 422.1] | 355.9 [212.5 to 596.2] | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 132.8 [96.16 to 183.4] | 247.1 [149.4 to 410.7] | 475.9 [128.0 to 1769] | 293.4 [141.6 to 607.7]

21. Secondary Outcome: Accumulation Ratio (Racc) for AUCtau of SAR245409: Day 15
Description: Accumulation ratio (Racc) for AUCtau, calculated as Day 15 dosing interval AUCtau divided by Day 1 dosing interval AUCtau.
Time Frame: as for outcome 3
Population: The PK analysis set. Here "N" signifies number of participant analyzed for this outcome measure and "n" signifies the number of subjects evaluable at the specific time points.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Groups:
- SAR245409 50mg Twice Daily: SAR245409 capsule administered twice, orally, at a dose of 50 mg on Day 1 of 21 day cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject.
Arm/Group | SAR245409 30mg | SAR245409 50mg | SAR245409 70mg | SAR245409 90mg | SAR245409 30mg Twice Daily | SAR245409 50mg Twice Daily | TNBC: SAR245409 70mg Once Daily | NSCLC: SAR245409 70mg Once Daily | CRC: SAR245409 70mg Once Daily | MEL: SAR245409 70mg Once Daily
Number analyzed (Participants) | 6 | 8 | 25 | 1 | 1 | 3 | 15 | 17 | 10 | 13
ratio | 1.189 [0.6118 to 2.311] | 1.004 [0.4637 to 2.175] | 0.9450 [0.6749 to 1.323] | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 1.800 [0.1724 to 18.79] | 1.256 [0.9407 to 1.676] | 0.9887 [0.7202 to 1.357] | 1.187 [0.7614 to 1.850] | 1.022 [0.6346 to 1.645]

22. Secondary Outcome: Accumulation Ratio (Racc) for Cmax of SAR245409: Day 15
Description: Accumulation ratio (Racc) for Cmax, calculated as Day 15 Cmax divided by Day 1 Cmax.
Time Frame: as for outcome 3
Population: as for outcome 21
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | SAR245409 30mg | SAR245409 50mg | SAR245409 70mg | SAR245409 90mg | SAR245409 30mg Twice Daily | SAR245409 50mg Twice Daily | TNBC: SAR245409 70mg Once Daily | NSCLC: SAR245409 70mg Once Daily | CRC: SAR245409 70mg Once Daily | MEL: SAR245409 70mg Once Daily
Number analyzed (Participants) | 6 | 8 | 25 | 1 | 1 | 3 | 17 | 17 | 10 | 13
Ratio | 1.041 [0.6293 to 1.722] | 0.8133 [0.3484 to 1.898] | 0.8962 [0.6151 to 1.306] | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | NA [NA to NA] — Data was not estimable if evaluable subjects were less than 3 as per the planned decision because only 2 collected values were not sufficient to calculate a reliable estimation. | 1.336 [0.03347 to 53.32] | 1.070 [0.8319 to 1.375] | 0.8950 [0.6951 to 1.152] | 0.9611 [0.6441 to 1.434] | 0.9942 [0.5447 to 1.815]

23. Secondary Outcome: pS6 Concentrations in Peripheral Blood Mononuclear Cells (PBMCs)
Description: pS6 Concentrations in PBMCs was measured during DDI Evaluation period and Cycle 1 for DE cohorts. DDI evaluation period is a 4-day period that was performed within 1 week prior to Day 1 Cycle 1. In DDI evaluation period, On Day 1, SAR245409 was be administered alone, and on Day 3, Pimasertib was administered alone. No data were planned to be collected for "Pimasertib (MSC1936369B) 60mg and SAR245409 30mg Twice Daily", "Pimasertib (MSC1936369B) 45mg and SAR245409 50mg Twice Daily", "Pimasertib (MSC1936369) 30mg and SAR245409 70mg Once Daily" and "Pimasertib (MSC1936369B) 60mg and SAR245409 90mg Once Daily" reporting arms.
Time Frame: DDI Evaluation: Day 1 and 3 (predose, 2, 4, 8 and 24 hours (hr) postdose); Day 2 and 4 (24 hr postdose); Cycle 1 Day 1 (C1D1) and C1D15 (predose, 2, 4, 8, 24 hr postdose); C1D2 and C1D16 (24 hr postdose); C1D19 (predose, 2 hr postdose)
Population: The Biomarker Analysis Set for pharmacodynamics (PD) marker analysis in PBMC included all subjects who received at least the first dose of both drugs and had provided at least one pre-dose sample and one post-dose sample. Here "n" signifies the number of subjects evaluable at the specific time points.
Measure: Mean (Standard Deviation); unit: fluorescence intensity
Groups:
- Pimasertib (MSC1936369B) 15mg and SAR245409 30mg Once Daily: Pimasertib (MSC1936369B) capsule was administered at a single oral dose of 15 milligram (mg) along with single oral dose of 30 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject.
- Pimasertib (MSC1936369B) 30mg and SAR245409 30mg Once Daily: Pimasertib (MSC1936369B) capsule was administered at a single oral dose of 30 mg along with single oral dose of 30 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject.
- Pimasertib (MSC1936369B) 15mg and SAR245409 50mg Once Daily: Pimasertib (MSC1936369B) capsule was administered at a single oral dose of 15 mg along with single oral dose of 50 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject.
- Pimasertib (MSC1936369B) 30mg and SAR245409 50mg Once Daily: Pimasertib (MSC1936369B) capsule was administered at a single oral dose of 30 mg along with single oral dose of 50 mg SAR245409 capsule on Day 1 of each 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject.
- Pimasertib (MSC1936369B) 60mg and SAR245409 50mg Once Daily: Pimasertib (MSC1936369B) capsule was administered at a single oral dose of 60 mg along with single oral dose of 50 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject
- Pimasertib (MSC1936369B) 60mg and SAR245409 70mg Once Daily: Pimasertib (MSC1936369B) capsule was administered at a single oral dose of 60 mg along with single oral dose of 70 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject.
- Pimasertib (MSC1936369B) 90mg and SAR245409 70mg Once Daily: Pimasertib (MSC1936369B) capsule was administered at a single oral dose of 90 mg along with single oral dose of 70 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject.
Arm/Group | Pimasertib (MSC1936369B) 15mg and SAR245409 30mg Once Daily | Pimasertib (MSC1936369B) 30mg and SAR245409 30mg Once Daily | Pimasertib (MSC1936369B) 15mg and SAR245409 50mg Once Daily | Pimasertib (MSC1936369B) 30mg and SAR245409 50mg Once Daily | Pimasertib (MSC1936369B) 60mg and SAR245409 50mg Once Daily | Pimasertib (MSC1936369B) 60mg and SAR245409 70mg Once Daily | Pimasertib (MSC1936369B) 90mg and SAR245409 70mg Once Daily
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 3 | 1
fluorescence intensity
  DDI Day 1: Pre-dose (n= 1, 0, 0, 0, 0, 0, 1) | 61.02 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 33.78 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  DDI Day 1: 2hr post-dose (n= 1,0,0,0,0,0,1) | 36.15 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 29.84 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  DDI Day 1: 4hr post-dose (n= 1,0,0,0,0,0,1) | 89.14 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 30.28 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  DDI Day 1: 8 hr post-dose(n= 1, 0, 0, 0, 0, 0, 1) | 54.54 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 44.88 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  DDI Day 1: 24hr post-dose (n= 1,0,0,0,0,0,0) | 88.80 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point.
  DDI Day 2: 24hr post-dose (n= 0,0,0,0,0,0,1) | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 28.86 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  DDI Day 3: Pre-dose (n= 1, 0, 0, 0, 0, 0, 1) | 57.51 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 14.90 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  DDI Day 3: 2hr post-dose (n= 1,0,0,0,0,0,1) | 55.93 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 34.06 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  DDI Day 3: 4hr post-dose (n= 1,0,0,0,0,0,1) | 36.76 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 1.03 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  DDI: Day 3: 8 hr post-dose(n= 1, 0, 0, 0, 0, 0, 1) | 1.08 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 40.40 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  DDI:Day 3: 24hr post-dose (n= 1,0,0,0,0,0,0) | 87.60 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point.
  DDI Day 4: 24hr post-dose (n= 0,0,0,0,0,0,1) | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 1.04 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  C1D1: Pre dose (n= 1,1,1,1,1,1,1) | 51.32 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 83.52 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 96.98 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 47.09 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 50.17 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 4.18 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 36.03 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  C1D1: 2hr postdose (n= 1,1,1,1,1,1,1) | 31.08 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 24.48 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 56.41 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 23.89 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 5.72 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 0.92 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.04 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  C1D1: 4hr postdose (n= 1,1,1,1,1,1,1) | 25.71 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 46.95 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 50.11 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 29.85 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 18.21 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 0.72 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 0.94 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  C1D1: 8hr postdose (n= 1,1,1,1,1,1,1) | 3.02 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.28 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 84.57 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 19.75 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 6.21 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.18 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 0.96 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  C1D1: 24hr postdose(n= 1,1,1,1,0,0,0) | 46.16 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 72.14 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 74.15 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 53.47 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point.
  C1D2: 24hr postdose (n= 0,0,0,0,1,1,1) | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 24.66 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.61 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.00 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  C1D15: pre-dose (n= 1,1,1,1,1,0,1) | 43.48 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 81.29 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 67.69 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.20 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 33.43 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 0.98 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  C1D15: 2hr postdose (n= 1,1,1,1,1,0,1) | 26.41 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 43.70 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 48.23 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 15.02 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 21.11 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 1.06 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  C1D15: 4hr postdose (n= 1,1,1,1,1,0,1) | 41.34 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 53.37 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 92.67 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 0.96 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 19.68 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 1.03 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  C1D15: 8hr postdose (n= 1,1,1,1,1,0,1) | 0.53 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 45.97 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 77.62 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 36.06 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 30.08 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 0.88 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  C1D15: 24hr postdose (n= 1,1,1,1,0,0,0) | 69.93 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 0.76 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 114.39 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 70.46 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point.
  C1D16: 24hr postdose (n= 0,0,0,0,1,0,1) | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 24.36 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 0.98 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  C1D19: pre-dose (n= 1,1,1,1,1,0,1) | 68.48 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 90.02 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 125.77 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 82.06 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 30.58 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 49.62 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  C1D19: 2hr postdose (n= 1,0,0,0,0,0,0) | 4.34 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point.

24. Secondary Outcome: pERK Concentrations in PBMCs
Description: pERK Concentrations in PBMCs was measured during DDI Evaluation period and Cycle 1 for DE cohorts. DDI evaluation period is a 4-day period that was performed within 1 week prior to Day 1 Cycle 1. In DDI evaluation period, On Day 1, SAR245409 was be administered alone, and on Day 3, Pimasertib was administered alone. No data were planned to be collected for "Pimasertib (MSC1936369B) 60mg and SAR245409 30mg Twice Daily", "Pimasertib (MSC1936369B) 45mg and SAR245409 50mg Twice Daily", "Pimasertib (MSC1936369) 30mg and SAR245409 70mg Once Daily" and "Pimasertib (MSC1936369B) 60mg and SAR245409 90mg Once Daily" reporting arms.
Time Frame: DDI Evaluation: Day 1 and 3 (predose, 2, 4, 8 and 24 hours (hr) postdose); Day 2 and 4 (24 hr postdose); C1D1 and C1D15 (predose, 2, 4, 8, 24 hr postdose); C1D2 and C1D16 (24 hr postdose); C1D19 (predose, 2 hr postdose)
Population: Biomarker Analysis Set for pharmacodynamics marker analysis in PBMC included all subjects who received at least first dose of both drugs and had provided at least one pre-dose sample and one post-dose sample. Here "N" signifies number of subject analysed for this outcome measure" and "n" signifies number of subject analysed at specific time point.
Measure: Mean (Standard Deviation); unit: fluorescence intensity
Arm/Group | Pimasertib (MSC1936369B) 15mg and SAR245409 30mg Once Daily | Pimasertib (MSC1936369B) 30mg and SAR245409 30mg Once Daily | Pimasertib (MSC1936369B) 15mg and SAR245409 50mg Once Daily | Pimasertib (MSC1936369B) 30mg and SAR245409 50mg Once Daily | Pimasertib (MSC1936369B) 60mg and SAR245409 50mg Once Daily | Pimasertib (MSC1936369B) 60mg and SAR245409 70mg Once Daily | Pimasertib (MSC1936369B) 90mg and SAR245409 70mg Once Daily
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 3 | 1
fluorescence intensity
  DDI Day 1: Predose (n= 1, 0, 0, 0, 0, 0, 1) | 6.77 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 10.55 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  DDI Day 1: 2 hr post-dose (n=1,0,0,0,0.0,1) | 8.74 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 10.17 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  DDI Day 1: 4 hr post-dose ((n=1,0,0,0,0,0,1) | 6.10 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 6.50 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  DDI Day 1: 8 hr post-dose(n= 1, 0, 0, 0, 0, 0, 1) | 7.42 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 9.36 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  DDI Day 1: 24 hr post-dose (n=1,0,0,0,0,0,0) | 10.84 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point.
  DDI Day 2: 24 hr post-dose ((n= 0,0,0,0,0,0,1) | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 8.32 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  DDI Day 3: Pre-dose (n= 1, 0, 0, 0, 0, 0, 1) | 9.46 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 8.94 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  DDI Day 3: 2 hr post-dose (n=1,0,0,0,0,0,1) | 3.12 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 15.82 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  DDI Day 3: 4 hr post-dose (n-1,0,0,0,0,0,1) | 6.74 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 0.68 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  DDI Day 3: 8 hr post-dose(n= 1, 0, 0, 0, 0, 0, 1) | 0.81 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 15.68 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  DDI Day 3: 24 hr post-dose (n=1,0,0,0,0,0,0) | 6.18 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point.
  DDI Day 4: 24 hr post-dose (n=0,0,0,0,0,0,1) | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 1.06 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  C1D1: Pre dose (n=1,1,1,1,1,1,1) | 5.56 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 3.45 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 6.96 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 3.25 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 3.35 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.97 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 7.42 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  C1D1: 2hr postdose(n= 1,1,1,1,1,1,1) | 2.37 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.33 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 2.78 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.54 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.40 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 0.95 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.04 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  C1D1: 4hr postdose(n= 1,1,1,1,1,1,1) | 2.85 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.37 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 2.91 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.24 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.96 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.11 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.01 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  C1D1: 8hr postdose(n= 1,1,1,1,1,1,1) | 0.67 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 0.94 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 3.40 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.96 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.27 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.12 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 0.82 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  C1D1: 24hr postdose(n= 1,1,1,1,0,0,0) | 6.23 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 2.15 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 4.59 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 6.26 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point.
  C1D2: 24hr postdose(n= 0,0,0,0,1,1,1) | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 3.45 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.26 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.05 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  C1D15: pre-dose(n= 1,1,1,1,1,0,1) | 3.79 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 2.26 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 5.29 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.41 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.93 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 2.03 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  C1D15: 2hr postdose (n= 1,1,1,1,1,0,1) | 2.16 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.34 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 2.83 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.60 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.55 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 0.94 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  C1D15: 4hr postdose (n= 1,1,1,1,1,0,1) | 1.87 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.34 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 2.50 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 0.94 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.20 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 0.81 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  C1D15: 8hr postdose (n= 1,1,1,1,1,0,1) | 1.92 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 2.08 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 3.38 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.10 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 1.74 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 0.99 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  C1D15: 24hr postdose (n= 1,1,1,1,0,0,0) | 4.97 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 0.94 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 5.33 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 4.70 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point.
  C1D16: 24hr postdose (n= 0,0,0,0,1,0,1) | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 2.36 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 0.99 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  C1D19: pre-dose (n= 1,1,1,1,1,0,1) | 6.54 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 2.61 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 4.47 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 5.44 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | 2.07 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | 5.72 (NA) — Data for standard deviation was not estimable as only one subject analyzed.
  C1D19: 2hr postdose (n= 1,0,0,0,0,0,0) | 1.60 (NA) — Data for standard deviation was not estimable as only one subject analyzed. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point. | NA (NA) — The parameter was not analyzed at specified time point because there were no subjects for which data was collected at the specified time point.

25. Secondary Outcome: Number of Subjects With Complete Tumor Response (CR), Partial Tumor Response (PR), or Stable Disease (SD)
Description: CR=Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeter (mm). PR=At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD=Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study. PD= At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From the date of randomisation every 6 weeks up to assessed up to 4 years
Population: The Efficacy Analysis Set (EEF) included all subjects who received at least 1 trial treatment dose (Pimasertib or SAR245409) and had radiographic baseline and at least one evaluable post baseline tumor assessment.
Measure: Number; unit: subjects
Groups:
- TNBC: Pimasertib 60mg and SAR245409 70mg Once Daily: Subjects with relapsed or refractory metastatic triple negative breast cancer (TNBC) defined as estrogen, progesterone, and human epidermal growth factor receptor 2 (HER2) negative carcinoma of the breast with no approved therapies in disease specific expansion (DSE) cohort received Pimasertib (MSC1936369B) capsule at a single oral dose of 60 mg along with single oral dose of 70 mg SAR245409 capsule on Day 1 of each 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DSE Cohort).
- NSCLC: Pimasertib 60mg and SAR245409 70mg Once Daily: Subjects with a histologically confirmed diagnosis of relapsed or refractory metastatic non-small cell lung cancer (NSCLC) in disease specific expansion (DSE) cohort received Pimasertib (MSC1936369B) capsule at a single oral dose of 60 mg along with single oral dose of 70 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DSE Cohort).
- CRC: Pimasertib 60mg and SAR245409 70mg Once Daily: Subjects with relapsed or refractory metastatic colorectal carcinoma/cancer (CRC) in DSE cohort received Pimasertib (MSC1936369B) capsule at a single oral dose of 60 mg along with single oral dose of 70 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DSE Cohort).
- MEL: Pimasertib 60mg and SAR245409 70mg Once Daily: Subjects with relapsed or refractory metastatic melanoma (MEL) in DSE cohort received Pimasertib (MSC1936369B) capsule at a single oral dose of 60 mg along with single oral dose of 70 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the subject (DSE Cohort).
Arm/Group | Pimasertib (MSC1936369B) 15mg and SAR245409 30mg Once Daily | Pimasertib (MSC1936369B) 30mg and SAR245409 30mg Once Daily | Pimasertib (MSC1936369B) 15mg and SAR245409 50mg Once Daily | Pimasertib (MSC1936369B) 30mg and SAR245409 50mg Once Daily | Pimasertib (MSC1936369B) 60mg and SAR245409 50mg Once Daily | Pimasertib (MSC1936369B) 30mg and SAR245409 70mg Once Daily | Pimasertib (MSC1936369B) 60mg and SAR245409 70mg Once Daily | Pimasertib (MSC1936369B) 90mg and SAR245409 70mg Once Daily | Pimasertib (MSC1936369B) 60mg and SAR245409 90mg Once Daily | Pimasertib (MSC1936369B) 60mg and SAR245409 30mg Twice Daily | Pimasertib (MSC1936369B) 45mg and SAR245409 50mg Twice Daily | TNBC: Pimasertib 60mg and SAR245409 70mg Once Daily | NSCLC: Pimasertib 60mg and SAR245409 70mg Once Daily | CRC: Pimasertib 60mg and SAR245409 70mg Once Daily | MEL: Pimasertib 60mg and SAR245409 70mg Once Daily
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 4 | 2 | 13 | 11 | 2 | 1 | 3 | 16 | 20 | 11 | 14
subjects
  Stable disease | 3 | 2 | 2 | 3 | 1 | 2 | 4 | 6 | 0 | 1 | 2 | 7 | 10 | 1 | 7
  Progressive disease | 0 | 0 | 1 | 1 | 1 | 0 | 9 | 3 | 2 | 0 | 1 | 8 | 6 | 9 | 4
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Partial Response | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Not Evaluable | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 1

ADVERSE EVENTS:
Time Frame: Baseline up to 30 Days after last dose; assessed up to 4 years
Groups:
- MSC1936369B (Pimasertib) 15mg and SAR245409 30mg Once Daily: MSC1936369B (Pimasertib) capsule administered at a single dose of 15 milligram (mg) on day 1 of each cycle (21 days) along with SAR245409 capsule administered at a single dose of 30 mg on day 1 of each cycle (21 days) (DE cohort).
- MSC1936369B (Pimasertib) 30mg and SAR245409 30mg Once Daily: MSC1936369B (Pimasertib) capsule administered at a single dose of 30 mg on day 1 of each cycle (21 days) along with SAR245409 capsule administered at a single dose of 30 mg on day 1 of each cycle (21 days) (DE cohort).
- MSC1936369B (Pimasertib) 15mg and SAR245409 50mg Once Daily: MSC1936369B (Pimasertib) capsule administered at a single dose of 15 mg on day 1 of each cycle (21 days) along with SAR245409 capsule administered at a single dose of 50 mg on day 1 of each cycle (21 days) (DE cohort).
- MSC1936369B (Pimasertib) 30mg and SAR245409 50mg Once Daily: MSC1936369B (Pimasertib) capsule administered at a single dose of 30 mg on day 1 of each cycle (21 days) along with SAR245409 capsule administered at a single dose of 50 mg on day 1 of each cycle (21 days) (DE cohort).
- MSC1936369B (Pimasertib) 60mg and SAR245409 50mg Once Daily: MSC1936369B (Pimasertib) capsule administered at a single dose of 60 mg on day 1 of each cycle (21 days) along with SAR245409 capsule administered at a single dose of 50 mg on day 1 of each cycle (21 days) (DE cohort).
- MSC1936369B (Pimasertib) 30mg and SAR245409 70mg Once Daily: MSC1936369B (Pimasertib) capsule administered at a single dose of 30 mg on day 1 of each cycle (21 days) along with SAR245409 capsule administered at a single dose of 70 mg on day 1 of each cycle (21 days) (DE cohort).
- MSC1936369B (Pimasertib) 60mg and SAR245409 70mg Once Daily: MSC1936369B (Pimasertib) capsule administered at a single dose of 60 mg on day 1 of each cycle (21 days) along with SAR245409 capsule administered at a single dose of 70 mg on day 1 of each cycle (21 days) (DE cohort).
- MSC1936369B (Pimasertib) 90mg and SAR245409 70mg Once Daily: MSC1936369B (Pimasertib) capsule administered at a single dose of 90 mg on day 1 of each cycle (21 days) along with SAR245409 capsule administered at a single dose of 70 mg on day 1 of each cycle (21 days) (DE cohort).
- MSC1936369B (Pimasertib) 60mg and SAR245409 90mg Once Daily: MSC1936369B (Pimasertib) capsule administered at a single dose of 60 mg on day 1 of each cycle (21 days) along with SAR245409 capsule administered at a single dose of 90 mg on day 1 of each cycle (21 days) (DE cohort).
- MSC1936369B (Pimasertib) 60mg and SAR245409 30mg Twice Daily: MSC1936369B (Pimasertib) capsule administered twice at a dose of 60 mg on day 1 and 15 of each cycle (21 days) along with SAR245409 capsule administered at a single dose of 30 mg on day 1 and 15 of each cycle (21 days) (DE cohort).
- MSC1936369B (Pimasertib) 45mg and SAR245409 50mg Twice Daily: MSC1936369B (Pimasertib) capsule administered twice at a dose of 45 mg on day 1 and 15 of each cycle (21 days) along with SAR245409 capsule administered at a single dose of 50 mg on day 1 and 15 of each cycle (21 days) (DE cohort).
- TNBC: Pimasertib 60mg and SAR245409 70mg Once Daily: Participants with relapsed or refractory metastatic triple negative breast cancer (TNBC) defined as estrogen, progesterone, and human epidermal growth factor receptor 2 (HER2) negative carcinoma of the breast with no approved therapies received Pimasertib (MSC1936369B) capsule at a single oral dose of 60 mg along with single oral dose of 70 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the participant (DSE Cohort).
- NSCLC: Pimasertib 60mg and SAR245409 70mg Once Daily: Participants with a histologically confirmed diagnosis of relapsed or refractory metastatic non-small cell lung cancer (NSCLC) in disease specific expansion (DSE) cohort received Pimasertib (MSC1936369B) capsule at a single oral dose of 60 mg along with single oral dose of 70 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the participant (DSE Cohort).
- CRC: Pimasertib 60mg and SAR245409 70mg Once Daily: Participants with relapsed or refractory metastatic colorectal carcinoma/cancer (CRC) in DSE cohort received Pimasertib (MSC1936369B) capsule at a single oral dose of 60 mg along with single oral dose of 70 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the participant (DSE Cohort).
- MEL: Pimasertib 60mg and SAR245409 70mg Once Daily: Participants with relapsed or refractory metastatic melanoma (MEL) in DSE cohort received Pimasertib (MSC1936369B) capsule at a single oral dose of 60 mg along with single oral dose of 70 mg SAR245409 capsule on Day 1 of 21 days cycle until disease progression, intolerable toxicity, Investigator's decision to discontinue treatment, or withdrawal of consent by the participant (DSE Cohort).
Arm/Group | MSC1936369B (Pimasertib) 15mg and SAR245409 30mg Once Daily | MSC1936369B (Pimasertib) 30mg and SAR245409 30mg Once Daily | MSC1936369B (Pimasertib) 15mg and SAR245409 50mg Once Daily | MSC1936369B (Pimasertib) 30mg and SAR245409 50mg Once Daily | MSC1936369B (Pimasertib) 60mg and SAR245409 50mg Once Daily | MSC1936369B (Pimasertib) 30mg and SAR245409 70mg Once Daily | MSC1936369B (Pimasertib) 60mg and SAR245409 70mg Once Daily | MSC1936369B (Pimasertib) 90mg and SAR245409 70mg Once Daily | MSC1936369B (Pimasertib) 60mg and SAR245409 90mg Once Daily | MSC1936369B (Pimasertib) 60mg and SAR245409 30mg Twice Daily | MSC1936369B (Pimasertib) 45mg and SAR245409 50mg Twice Daily | TNBC: Pimasertib 60mg and SAR245409 70mg Once Daily | NSCLC: Pimasertib 60mg and SAR245409 70mg Once Daily | CRC: Pimasertib 60mg and SAR245409 70mg Once Daily | MEL: Pimasertib 60mg and SAR245409 70mg Once Daily
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 2/3 | 1/4 | 1/4 | 1/3 | 14/19 | 10/14 | 1/3 | 2/3 | 3/4 | 16/26 | 13/24 | 10/18 | 8/15
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 4/4 | 4/4 | 3/3 | 19/19 | 14/14 | 3/3 | 3/3 | 4/4 | 26/26 | 24/24 | 18/18 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MSC1936369B (Pimasertib) 15mg and SAR245409 30mg Once Daily (N=3) | MSC1936369B (Pimasertib) 30mg and SAR245409 30mg Once Daily (N=3) | MSC1936369B (Pimasertib) 15mg and SAR245409 50mg Once Daily (N=3) | MSC1936369B (Pimasertib) 30mg and SAR245409 50mg Once Daily (N=4) | MSC1936369B (Pimasertib) 60mg and SAR245409 50mg Once Daily (N=4) | MSC1936369B (Pimasertib) 30mg and SAR245409 70mg Once Daily (N=3) | MSC1936369B (Pimasertib) 60mg and SAR245409 70mg Once Daily (N=19) | MSC1936369B (Pimasertib) 90mg and SAR245409 70mg Once Daily (N=14) | MSC1936369B (Pimasertib) 60mg and SAR245409 90mg Once Daily (N=3) | MSC1936369B (Pimasertib) 60mg and SAR245409 30mg Twice Daily (N=3) | MSC1936369B (Pimasertib) 45mg and SAR245409 50mg Twice Daily (N=4) | TNBC: Pimasertib 60mg and SAR245409 70mg Once Daily (N=26) | NSCLC: Pimasertib 60mg and SAR245409 70mg Once Daily (N=24) | CRC: Pimasertib 60mg and SAR245409 70mg Once Daily (N=18) | MEL: Pimasertib 60mg and SAR245409 70mg Once Daily (N=15)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 0
VOMITING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ASCITES (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0
DYSPHAGIA (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
PYREXIA (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 0 | 1 | 1 | 2 | 1 | 2 | 0
DISEASE PROGRESSION (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 2 | 1 | 3 | 2 | 0
GAIT DISTURBANCE (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HEPATIC FAILURE (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CELLULITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
FUNGAL SKIN INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INFLUENZA (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PELVIC ABSCESS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BLOOD CREATININE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LETHARGY (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PRESYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
HALLUCINATION (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
VULVOVAGINAL PAIN (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 2 | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DERMATITIS EXFOLIATIVE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
HYPERTENSION (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
HYPOTENSION (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0
FATIGUE (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
BILE DUCT STENOSIS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
LUNG INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
SUPERIOR VENA CAVA SYNDROME (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
TEMPORAL ARTERITIS (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
ATRIAL FLUTTER (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
BRADYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
RIGHT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
PANCREATITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
FATIGUE (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
GENERALISED OEDEMA (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 1
SEPSIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
ABDOMINAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ESCHERICHIA INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ESCHERICHIA SEPSIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
HEMIPARESIS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
EMBOLISM (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ANAPHYLACTIC REACTION (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MSC1936369B (Pimasertib) 15mg and SAR245409 30mg Once Daily (N=3) | MSC1936369B (Pimasertib) 30mg and SAR245409 30mg Once Daily (N=3) | MSC1936369B (Pimasertib) 15mg and SAR245409 50mg Once Daily (N=3) | MSC1936369B (Pimasertib) 30mg and SAR245409 50mg Once Daily (N=4) | MSC1936369B (Pimasertib) 60mg and SAR245409 50mg Once Daily (N=4) | MSC1936369B (Pimasertib) 30mg and SAR245409 70mg Once Daily (N=3) | MSC1936369B (Pimasertib) 60mg and SAR245409 70mg Once Daily (N=19) | MSC1936369B (Pimasertib) 90mg and SAR245409 70mg Once Daily (N=14) | MSC1936369B (Pimasertib) 60mg and SAR245409 90mg Once Daily (N=3) | MSC1936369B (Pimasertib) 60mg and SAR245409 30mg Twice Daily (N=3) | MSC1936369B (Pimasertib) 45mg and SAR245409 50mg Twice Daily (N=4) | TNBC: Pimasertib 60mg and SAR245409 70mg Once Daily (N=26) | NSCLC: Pimasertib 60mg and SAR245409 70mg Once Daily (N=24) | CRC: Pimasertib 60mg and SAR245409 70mg Once Daily (N=18) | MEL: Pimasertib 60mg and SAR245409 70mg Once Daily (N=15)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 2 | 1 | 1 | 0 | 7 | 3 | 1 | 0 | 0 | 4 | 2 | 4 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 5 | 0 | 1 | 0
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
ANAEMIA MACROCYTIC (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 0
SINUS TACHYCARDIA (Cardiac disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
PALPITATIONS (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ATRIAL FLUTTER (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
SINUS BRADYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
HEARING IMPAIRED (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
HYPOTHYROIDISM (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SUBRETINAL FLUID (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 4 | 5 | 0 | 0 | 0 | 1 | 2 | 0 | 0
VISUAL ACUITY REDUCED (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 3 | 0 | 0 | 0 | 6 | 6 | 2 | 2
VISUAL IMPAIRMENT (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 1 | 1 | 0 | 6 | 0 | 0 | 1
RETINAL DETACHMENT (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 1 | 1 | 0 | 3 | 8 | 5 | 3
PERIORBITAL OEDEMA (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1
VISION BLURRED (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 1 | 0 | 5 | 4 | 4 | 3
DETACHMENT OF RETINAL PIGMENT EPITHELIUM (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 0
MACULAR DETACHMENT (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 5 | 1 | 2 | 3
VITREOUS FLOATERS (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
PHOTOPSIA (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1
RETINAL HAEMORRHAGE (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BLEPHARITIS (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CATARACT (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CHORIORETINOPATHY (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DIPLOPIA (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1
DRY EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
EYE OEDEMA (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
EYE PAIN (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
GLAUCOMA (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MACULAR FIBROSIS (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MACULAR HOLE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
RETINAL EXUDATES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
XANTHOPSIA (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Halo Vision (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
EYE COLOUR CHANGE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
EYE DISCHARGE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
EYE PRURITUS (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
EYELID FUNCTION DISORDER (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
EYELIDS PRURITUS (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
METAMORPHOPSIA (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
RETINAL DEGENERATION (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 3 | 2 | 2 | 4 | 2 | 2 | 10 | 13 | 1 | 3 | 1 | 22 | 19 | 13 | 10
NAUSEA (Gastrointestinal disorders) | 1 | 2 | 2 | 1 | 1 | 3 | 7 | 8 | 2 | 3 | 0 | 11 | 15 | 8 | 7
VOMITING (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2 | 3 | 8 | 9 | 1 | 2 | 3 | 12 | 11 | 7 | 8
STOMATITIS (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 3 | 1 | 2 | 0 | 11 | 5 | 5 | 2
DRY MOUTH (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 2 | 1 | 1 | 2 | 3 | 2 | 4 | 2
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 1
DYSPEPSIA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 1 | 2 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 1 | 6 | 3 | 1 | 3
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 0 | 6 | 5 | 3 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FLATULENCE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GASTRITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ASCITES (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
DIVERTICULUM (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DYSPHAGIA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ERUCTATION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
HIATUS HERNIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
LIP ULCERATION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MELAENA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MOUTH ULCERATION (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OESOPHAGITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ORAL DYSAESTHESIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ORAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
REFLUX GASTRITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
RETCHING (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
SENSITIVITY OF TEETH (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TOOTHACHE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ENLARGED UVULA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
HYPOAESTHESIA ORAL (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ANAL FISSURE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
GASTROINTESTINAL INFLAMMATION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
GLOSSITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
NEUROGENIC BOWEL (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ORAL DISCOMFORT (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ORAL MUCOSAL ERYTHEMA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
FATIGUE (General disorders) | 3 | 1 | 2 | 2 | 3 | 2 | 8 | 9 | 2 | 3 | 4 | 17 | 14 | 9 | 4
OEDEMA PERIPHERAL (General disorders) | 1 | 2 | 3 | 1 | 1 | 0 | 7 | 7 | 1 | 2 | 1 | 7 | 5 | 3 | 4
PYREXIA (General disorders) | 2 | 1 | 0 | 0 | 1 | 1 | 5 | 4 | 1 | 1 | 0 | 7 | 2 | 5 | 4
ASTHENIA (General disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 2 | 0 | 4 | 2 | 3 | 3
CHILLS (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 0 | 1 | 2 | 4 | 2 | 0 | 2
FACE OEDEMA (General disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 3 | 0 | 1 | 1 | 3 | 2 | 2 | 1
CHEST DISCOMFORT (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
CHEST PAIN (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
GAIT DISTURBANCE (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
HERNIA PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LOCAL SWELLING (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MALAISE (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
MUCOSAL INFLAMMATION (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
PAIN (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0
PERIPHERAL SWELLING (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
THROMBOSIS IN DEVICE (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FACIAL PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
GENERALISED OEDEMA (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 2
PERFORMANCE STATUS DECREASED (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
EARLY SATIETY (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
INFLAMMATION (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
MUCOSAL DRYNESS (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
NODULE (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
TEMPERATURE INTOLERANCE (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
JAUNDICE (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
HEPATITIS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
PORTAL HYPERTENSION (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 0 | 0 | 0 | 2 | 0 | 3 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0
CELLULITIS (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
BACTERIAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
BODY TINEA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BRONCHITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ENTEROCOCCAL BACTERAEMIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FUNGAL SKIN INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LUNG INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OESOPHAGEAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ORAL FUNGAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
RASH PUSTULAR (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
SINUSITIS BACTERIAL (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SKIN INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TINEA CRURIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
WOUND INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ORAL CANDIDIASIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
DEVICE RELATED INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
ORAL HERPES (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
PARONYCHIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
RASH PUSTULAR (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
BACTERIAL VAGINOSIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
CATHETER SITE INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
FURUNCLE (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HERPES VIRUS INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
LARYNGITIS VIRAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
LOCALISED INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
NAIL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ORAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
PNEUMONIA FUNGAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
VAGINAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INCISION SITE ERYTHEMA (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 5 | 1 | 0 | 1 | 1 | 2 | 2 | 0
BLOOD CREATININE INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 1 | 1 | 1 | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 1 | 1 | 1 | 1 | 0
EJECTION FRACTION DECREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 2 | 2 | 3 | 0 | 2
WEIGHT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 0
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 0
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 2 | 2 | 1
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 3 | 3 | 0
BLOOD CHOLESTEROL INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 6 | 5 | 4 | 4
BLOOD POTASSIUM DECREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BLOOD UREA INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BLOOD URINE PRESENT (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HAEMOGLOBIN DECREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
INTRAOCULAR PRESSURE INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PLATELET COUNT DECREASED (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
URINE OUTPUT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
WEIGHT INCREASED (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
HEART RATE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
VITAMIN D DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
BLOOD PRESSURE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
BLOOD TESTOSTERONE DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
BREATH SOUNDS ABNORMAL (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
LIPASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
PROTHROMBIN TIME PROLONGED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
TRANSAMINASES INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
TROPONIN INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 1 | 2 | 6 | 5 | 1 | 2 | 0 | 8 | 7 | 4 | 5
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 6 | 2 | 0 | 1 | 0 | 9 | 1 | 2 | 2
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 3 | 1 | 2 | 2 | 0 | 6 | 1 | 4 | 2
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 2 | 1 | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 1 | 1 | 0 | 1 | 1 | 1 | 3 | 0
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 1 | 0 | 5 | 1 | 4 | 0
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 1 | 0 | 3 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 4 | 1
FLUID RETENTION (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
FLUID OVERLOAD (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
HYPERAMYLASAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
MALNUTRITION (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 1 | 0 | 2 | 3 | 0 | 4
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 2 | 4 | 1 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 2 | 1 | 3
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
JOINT EFFUSION (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 3 | 0 | 1
MUSCULOSKELETAL CHEST PAIN (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 2
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
MUSCLE TWITCHING (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ACROCHORDON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
INFECTED NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ONCOLOGIC COMPLICATION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
DIZZINESS (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 2 | 0 | 0 | 0 | 7 | 9 | 1 | 3
HEADACHE (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 2 | 1 | 4 | 6 | 2 | 3
DYSGEUSIA (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 3
SOMNOLENCE (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0
COGNITIVE DISORDER (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 1
PRESYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
TREMOR (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
ATAXIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
BRAIN OEDEMA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DIZZINESS EXERTIONAL (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HEMIANOPIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPOAESTHESIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
LETHARGY (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
MEMORY IMPAIRMENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
PARAESTHESIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
PERONEAL NERVE PALSY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SPINAL CORD COMPRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
TRANSVERSE SINUS THROMBOSIS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
VISUAL FIELD DEFECT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
BALANCE DISORDER (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
PARAPLEGIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
BURNING SENSATION (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
DYSARTHRIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPOKINESIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
NEURALGIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SCIATICA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
SINUS HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ANXIETY (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 4 | 3 | 2 | 3
INSOMNIA (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 4 | 0 | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0
AGITATION (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
DEPRESSED MOOD (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DEPRESSION (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
DEPRESSIVE SYMPTOM (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
DELIRIUM (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
MAJOR DEPRESSION (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
MENTAL STATUS CHANGES (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
HAEMATURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
DYSURIA (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1
NOCTURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PROTEINURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
URINARY RETENTION (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
CHROMATURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
MICTURITION URGENCY (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
NEUROGENIC BLADDER (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
POLYURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
URINARY INCONTINENCE (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
URINARY TRACT PAIN (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0
BREAST PAIN (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PELVIC PAIN (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BREAST MASS (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 4 | 5 | 0 | 1 | 1 | 4 | 6 | 1 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 3 | 0 | 1 | 2 | 0 | 1 | 0 | 3 | 4 | 2 | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 2 | 4 | 2 | 1
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 2
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 2
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 2 | 1
SPUTUM INCREASED (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TACHYPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
LARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 2 | 0 | 2 | 9 | 6 | 1 | 2 | 1 | 13 | 8 | 4 | 7
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2 | 3 | 0 | 6 | 5 | 1 | 2 | 3 | 6 | 12 | 4 | 5
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 2 | 0 | 2 | 3 | 0 | 0 | 0 | 5 | 5 | 1 | 5
RASH (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 2 | 2 | 0 | 3
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 2 | 2 | 0 | 3
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
SKIN DISORDER (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ACNE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DERMATITIS EXFOLIATIVE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
GENERALISED ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HAIR COLOUR CHANGES (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HAIR GROWTH ABNORMAL (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HYPERHIDROSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
PETECHIAE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SKIN BURNING SENSATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 1
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
NAIL DISCOLOURATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPERTENSION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 0 | 1 | 3 | 3 | 1 | 5
DEEP VEIN THROMBOSIS (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
FLUSHING (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HOT FLUSH (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HYPOTENSION (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 2 | 0 | 1
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
SUPERIOR VENA CAVA SYNDROME (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
CAPILLARY LEAK SYNDROME (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
LYMPHOEDEMA (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
PHLEBITIS SUPERFICIAL (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other